CLINICAL TRIAL: NCT07176091
Title: Transcranial Direct Current Stimulation Combined With Transcranial Magnetic Stimulation for Motor and Non-Motor Symptoms of Parkinsonian Syndromes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Cheng-Jie Mao, Associate Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LK2025027
Record Dates: First submitted 2025-08-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Parkinsonism; Transcranial Direct Current Stimulation; Transcranial Magnetic Stimilation; Intermittent Theta Burst Stimulation; Primary Motor Cortex
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined treatment of tDCS and TMS (Experimental): Bilateral pre-treatment with tDCS is carried out for 10 minutes. The current is 2 mA, and the electrodes are spaced 5 cm apart. The current gradually rises and falls in the first and last 30 seconds. Subsequently, the bilateral primary motor cortex (M1 area) of the patient is stimulated with iTBS at a frequency of 5 Hz. The magnetic field intensity is set at 80% of the resting motor threshold. Each train contains 10 pulses, and each pulse consists of 3 bidirectional pulses at 50 Hz. The interval between each train is 8 seconds. There are 60 trains per session (1800 pulses per session), and the treatment lasts for 5 days in total.
  Interventions: Device: Combined treatment of tDCS and rTMS
- sham-tDCS combined with real TMS (Active Comparator): Participants received sham transcranial direct current stimulation combined with intermittent theta burst stimulation for a total of 5 days
  Interventions: Device: sham-tDCS combined with real TMS

INTERVENTIONS:
Device: Combined treatment of tDCS and rTMS — Bilateral pre-treatment with tDCS is carried out for 10 minutes. The current is 2 mA, and the electrodes are spaced 5 cm apart. The current gradually rises and falls in the first and last 30 seconds. Subsequently, the bilateral primary motor cortex (M1 area) of the patient is stimulated with iTBS at a frequency of 5 Hz. The magnetic field intensity is set at 80% of the resting motor threshold. Each train contains 10 pulses, and each pulse consists of 3 bidirectional pulses at 50 Hz. The interval between each train is 8 seconds. There are 60 trains per session (1800 pulses per session), and the treatment lasts for 5 days in total.
  Other Names: The group treated with tDCS; The group treated with rTMS
  Arms: Combined treatment of tDCS and TMS
Device: sham-tDCS combined with real TMS — Participants received sham transcranial direct current stimulation combined with intermittent theta burst stimulation for a total of 5 days
  Arms: sham-tDCS combined with real TMS

SUMMARY:
The combination of transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS) is an increasingly recognized neuromodulation strategy in the treatment of Parkinsonian syndromes, showing particular potential in improving both motor and non-motor symptoms. Typical motor symptoms such as bradykinesia, rigidity, and tremor, along with various non-motor symptoms including pain, depression, and fatigue, collectively contribute to the major burden of the disease. tDCS modulates cortical excitability via weak electrical currents, while TMS induces neuronal depolarization using time-varying magnetic fields. Their combined application allows synergistic multi-target intervention on the motor cortex and related neural networks. However, high-quality randomized controlled trials focusing on the combined tDCS-TMS approach in Parkinsonian syndromes remain relatively limited, and its long-term efficacy and underlying mechanisms have not yet been systematically established.Beyond systematically evaluating the efficacy and safety of combined tDCS-TMS on motor and non-motor functions in patients with Parkinsonian syndromes, this study also aims to integrate multimodal neuroimaging and neurophysiological techniques to investigate the key mechanisms by which the combined modulation acts on basal ganglia-cortical circuits and the default mode network. Furthermore, we will analyze the specificity and synergism of its effects across different symptomatic domains.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder caused by the degeneration of dopaminergic neurons, with pathological mechanisms involving abnormal activity in neural networks. tDCS modulates the excitability of cortical neurons via weak electrical currents, while TMS stimulates specific brain regions using magnetic fields. Both techniques are capable of regulating brain network activity. Their combined application may enable more comprehensive modulation of pathological neural networks and theoretically produce synergistic improvements across multiple symptoms of Parkinson's disease.Parkinsonian syndromes are characterized not only by motor symptoms but also by non-motor manifestations such as cognitive impairment, depression, and sleep disturbances. The combination of tDCS and TMS may not only enhance the effects of each technique applied alone but also allow simultaneous multi-target interventions, leading to more holistic symptom management.Although research on combined tDCS-TMS in Parkinsonian syndromes remains limited, evidence from related fields supports the feasibility and potential benefits of such neuromodulatory strategies. This study employs a randomized, double-blind design to evaluate the efficacy and safety of combined tDCS-TMS treatment in patients with Parkinsonian syndromes. By using single-pulse resting-state EEG and functional magnetic resonance imaging (fMRI), we aim to directly capture changes in cortical activity mechanisms within the M1 region before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ① The diagnosis of primary Parkinson's disease conforms to the clinical diagnostic criteria for PD established by the Movement Disorders Society (MDS) in 2015.

  * The diagnosis of Parkinson's plus syndromes conforms to the following: The diagnosis of multiple system atrophy conforms to the clinical diagnostic criteria for MSA established by the MDS in 2022; the diagnosis of progressive supranuclear palsy conforms to the clinical diagnostic criteria for PSP established by the MDS in 2017.

    * Having one or more of the following conditions: Complicating with one or more sleep disorders; Complicating with cognitive impairment, with a Mini-Mental State Examination (MMSE) score < 27 points and/or a Montreal Cognitive Assessment (MoCA) score < 26 points; Complicating with freezing of gait; Accompanied by one or more types of PD pain, with a Numerical Rating Scale (NRS) score ≥ 3 points and lasting for 3 months or more.

      * The medications for treating PD have been stably used for more than 2 weeks, and the original medication treatment regimen is maintained during the transcranial magnetic stimulation (TMS) treatment period.

        * Analgesic medications such as non-steroidal anti-inflammatory drugs have been stably used for more than 16 weeks, and the original treatment dosage is maintained unchanged during the trial period.

          ⑥ There is no obvious atrophy and no other characteristic changes in the head CT/MRI examination.

          ⑦ The patient and their family members have been informed of the examination items to be carried out, have given their informed consent, and have signed the informed consent form.

Exclusion Criteria:

* ① Patients with other diseases that may affect the sensation of peripheral nerves, including diabetes mellitus, herpes infection, long-term use of specific medications or excessive alcohol consumption, stroke, spinal cord lesions, etc.;

  * Patients complicated with severe depression or mental disorders;

    * Patients with severe cognitive impairment, with a Mini-Mental State Examination (MMSE) score and/or a Montreal Cognitive Assessment (MoCA) score ≤ 9 points; ④ Patients complicated with intracranial organic lesions or craniocerebral trauma; ⑤ Patients complicated with severe organic lesions of the heart, liver, kidney, etc.; ⑥ Patients who cannot complete head MRI examination, transcranial direct current stimulation (tDCS) or transcranial magnetic stimulation (TMS) treatment due to claustrophobia, having implanted devices such as a pacemaker in the body, a history of epilepsy, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment with the KPPS | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  King's PD Pain Scale (KPPS) includes 14 items rating the severity and frequency of pain, each item scored by severity (0-3) multiplied by frequency (0-4), resulting in a subscore of 0 to 12, with a total possible score range from 0 to 168. Higher scores indicate greater symptom severities and more serious influence.
Assessment with the MKPPS | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  Modified King's PD Pain Scale (MKPPS)，the modified version which is more suitable for Chinese people, combined with Ford's pain subtypes basing on the original. It covers five main domains, including 16 items, each item scored by severity (0-3) multiplied by frequency (0-4), resulting in a total possible score range from 0 to 192. Higher scores indicate greater symptom severities and more serious influence.
Change in Pain Intensity Scores (VAS) | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  VAS, a 0-10 numeric rating scale with 0= no pain and 10=maximal pain. Higher scores indicate greater symptom severities and more serious influence.

SECONDARY OUTCOMES:
Changes in MDS-UPDRS I | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The participants will be evaluated in their "ON" medication states. The scales used to assess non-motor symptoms included parts I (ranging from 0 to 52) and II (ranging from 0 to 52) of the MDS-UPDRS, with higher scores indicating more severe symptoms
Change in MDS-UPDRS II | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The participants will be evaluated in their "ON" medication states. The scales used to assess non-motor symptoms included parts I (ranging from 0 to 52) and II (ranging from 0 to 52) of the MDS-UPDRS, with higher scores indicating more severe symptoms.
Change in MDS-UPDRS III | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The participants will be evaluated in their "ON" medication states. The scales used to assess motor symptoms included parts III (ranging from 0 to 132) and IV (ranging from 0 to 24) of the MDS-UPDRS, with higher scores indicating more severe symptoms.
Changes in PD Depression Score | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The depression score (ranging from 0 to 76 with higher scores indicating more severe depression) from the 24 items Hamilton Depression Scale (HAMD).
Changes in PD Anxiety Score | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The anxiety score (ranging from 0 to 60 with higher scores indicating more severe anxiety) from the 14 items Hamilton Anxiety Scale (HAMA).
Changes in PD Autonomic Symptoms Score | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The Scale for Outcomes in Parkinson's disease for Autonomic Symptoms (SCOUP-AUT, maximal score 67, with higher scores indicating higher autonomic nervous system dysfunction).
Changes in PD Sleep Problem Score | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The sleep problem index (from 0 to 68 with higher scores indicating more severe sleep problem) from the PD Sleep Scale-2 (PDSS-2).
Changes in PD Daytime Sleepiness Score | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  The daytime sleepiness will be assessed by the Epworth Sleeping Scale (ESS), maximal score 24, with higher scores indicating more severe symptoms.
Changes in PD Quality of Life Score | at baseline, on day 1 after treatment, and at 1 month and 3 months after treatment
  We will also assess change in quality of life from the Parkinson's Disease Questionnaire-39 (PDQ-39), ranging from 0 to 156 with higher scores indicating more serious influence.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No